CLINICAL TRIAL: NCT04773652
Title: Predictors of Adverse Left Ventricular Remodeling and Final Infarct Size After Primary Percutaneous Coronary Intervention for ST Elevation Myocardial Infarction: A Strain Analysis Study Using Echocardiography and Feature Tracking Cardiac Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Aswan Heart Centre (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Cardiology consultant, Cairo University
Other Study IDs: R-4-2020
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: ST Elevation Myocardial Infarction; Remodeling, Left Ventricle
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: speckle tracking echo — Two-dimensional and 3D Speckle tracking echocardiography and feature tracking CMR will be performed twice: within 48 hours of admission and 3 months following the index event.
  Other Names: Feature tracking CMR

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) is one of the most important causes of death and disability around the world.

The main goal in the management of acute myocardial infarction (AMI) is early restoration of coronary artery flow in order to preserve viable myocardium. Primary percutaneous coronary intervention (PCI) has proven to be superior to other reperfusion strategies in terms of mortality reduction and preservation of left ventricular (LV) function. Despite improvements in the treatment of MI, 30% of patients show LV remodeling post-MI. Over time, remodeling adversely affects cardiac function and can lead to significant morbidity and mortality. Early risk stratification is essential to identify patients who will benefit from close follow-up and intense medical therapy.

The most widely investigated functional left ventricular (LV) characteristic to predict patient outcome after STEMI is LV ejection fraction (LVEF). Several structural LV characteristics have also shown to be important predictors of cardiovascular adverse events and death, including LV end diastolic volume (LVEDV), end systolic volume (LVESV) and mass (LVM).

Cardiovascular magnetic resonance (CMR) imaging is the current reference standard for assessing ventricular volumes and mass. Adverse remodeling results from an inability of the heart to maintain geometry post MI in the context of large infarcts and increased wall stresses.

The compensatory hypertrophic response of the remote non-infarcted myocardium (end diastolic wall thickness (EDWT) and end systolic wall thickness (ESWT)) might also play an important role in the remodeling after myocardial infarction but this needs to be investigated.

Infarct size -as a crucial endpoint for adverse remodeling- is influenced by several factors: - the size of the area at risk (AAR) (myocardium supplied by the culprit vessel); residual flow to the ischemic territory (e.g., collateral flow); myocardial metabolic demand; and the duration of coronary occlusion.

Assessment of the size and distribution of the infarction area after revascularization therapy can facilitate prompt and appropriate clinical intervention. Biomarkers such as troponin and creatine kinase are mainly used for AMI identification but lack myocardial specificity and may overestimate the (IS). Left ventricle ejection fraction (LVEF) fails to detect minimal and early pathological changes. The myocardial damage following STEMI can be assessed accurately by delayed gadolinium enhancement imaging using CMR imaging. In the acute phase of a STEMI, the extracellular space is increased in the infarct region due to a combination of necrosis, hemorrhage, and edema. The extent of hyper enhancement in the acute phase has been related to the outcome in patients with STEMI. However, later on the necrotic tissue is replaced by fibrotic scar tissue also with increased extracellular space. This process leads to ongoing 'infarct shrinkage' after the first week until the infarction reaches its final size after ∼30 days. - - Measurement of hyper enhancement in the acute phase of an infarction might therefore overestimate the necrotic infarct size, whereas 'final extent of hyper enhancement' is more precisely related to the amount of necrotic tissue. In STEMI patients the prognostic importance and predictors of the final infarct size are not fully elucidated.

Myocardial strain is a quantitative index based on measuring myocardial deformation during a cardiac cycle. Major tools for detecting changes in myocardial strain include CMR tagging, CMR feature tracking (FT-CMR) and speckle tracking echocardiography (STE). Previous studies have shown an advantage of strain in sensitively and accurately diagnosing and assessing IS compared to traditional functional indexes. However, the degree to which strain analysis can reflect the infarction areas quantified by CMR, adverse LV remodeling as well as the diagnostic accuracy of this analysis is still under dispute. In the past 3 years in particular, newly developed three-dimensional (3D) STE has overcome the inherent shortcomings of two-dimensional (2D) STE.

DETAILED DESCRIPTION:
The study will enroll 100 consecutive patients with acute STEMI presenting to Aswan Heart Centre catheterization-lab for primary PCI matching the selection criteria. Diagnosis of STEMI will be based upon:

Sustained ST-segment elevation of at least 1 mm in at least 2 contiguous leads or new/presumably new left bundle branch block, plus

* Typical anginal pain
* or diagnostic levels of serum cardiac biomarkers
* or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

The study patients will undergo primary PCI according to the recent practice guidelines and the local hospital policy in managing ST elevation MI patients. Echocardiography and CMR will be performed twice: within 48 hours of admission and 3 months following the index event.

Management

* Twelve-lead electrocardiogram will be recorded at baseline and 30-min post-procedure. The ST-segment changes will be evaluated in the single lead with the most prominent ST-segment elevation before intervention. The ST-segment elevation will be measured to the nearest 0.5 mm at 60 ms after the J point. Significant ST segment resolution (STR) is defined as a reduction in ST-segment elevation of 50% after 30 min of infarct artery recanalization .
* Immediately before the procedure, patients will receive aspirin (300 mg), clopidogrel (600 mg), or ticagrelor (180 mg). Adjunctive pharmacological treatment during the procedure will include:

  1. Unfractionated heparin as an initial bolus of 70 U/kg and additional boluses during the procedure to achieve an activated clotting time of 250 to 350 s (200 to 250 s if Glycoprotein IIb/IIIa (GPIIb/IIIa) antagonist is used). Heparin will be discontinued at the end of percutaneous coronary intervention.
  2. The use of a GPIIb/IIIa antagonist during the procedure, primary PCI technique, indications, and methods of thrombectomy if indicated will be done under the regulations of the local hospital policy and the most recent practice guidelines.

The following data will be collected:

1. Clinical data:

   These include age, gender, weight, height, body mass index, body surface area, smoking status, history of hypertension or diabetes mellitus, dyslipidemia, prior history of coronary artery disease (CAD), and previous coronary interventions. Times from onset of pain to first medical contact, to definitive diagnosis, to needle and to restoration of coronary flow will be recorded as well.
2. Laboratory work up:

   Complete blood count, INR, cardiac biomarkers (total CK, CK-MB, troponin), Brain natriuretic peptide (BNP), soluble suppression of tumorigenicity 2 (sST2), liver enzymes (ALT and AST), urea and creatinine, and serum electrolytes (Na, K).
3. Angiographic data:

   * The thrombolysis in myocardial infarction (TIMI) flow grade:

TIMI flow grade will be assessed at three different time points; immediately after the diagnostic coronary angiography, after wiring the culprit vessel and at the end of the procedure.

* TIMI 0 flow: refers to the absence of any antegrade flow beyond a coronary occlusion.
* TIMI 1 flow: refers to faint antegrade coronary flow beyond the occlusion, with incomplete filling of the distal coronary bed.
* TIMI 2 flow: refers to delayed or sluggish antegrade flow with complete filling of the distal territory.
* TIMI 3 flow: refers to normal antegrade flow with complete filling of the distal territory.

  • The myocardial blush grade (MBG): Myocardial blush grade evaluates contrast density in the myocardial region of the infarct-related artery compared to regions of non-infarct-related arteries on coronary angiography. It will be reported at the end of the procedure.
* MBG 0: no myocardial blush.
* MBG 1: minimal myocardial blush or contrast density.
* MBG 2: moderate blush or contrast density, but less than a contralateral or ipsilateral non infarct-related artery.
* MBG 3: normal myocardial blush or contrast density similar to a contralateral or ipsilateral non infarct-related artery.

When myocardial blush persisted ("staining"), this phenomenon suggested leakage of the contrast medium into the extravascular space, and will be graded 0 Angiographic incomplete reperfusion is defined as TIMI flow grade < 2 or MBG < 2.

Echocardiography protocol:

Patients will undergo transthoracic echocardiography using xMATRIX X5-1 phased array sector probe (1 - 5 MHz) of the Philips iE33 xMATRIX and EPIQ 7 machines (Philips Medical Systems, Andover, MA, USA). The blood pressure and heart rate during the study will be recorded.

1. Conventional echocardiography:

   Standard views will be obtained and analyzed in accordance with the American Society of Echocardiography guidelines. . The following variables will be noted:
   1. Left ventricular ejection fraction: calculated by the modified Simpson's rule by tracing the endocardial border at end-diastole and end-systole in the two-chamber and four-chamber views.
   2. Left ventricular end-diastolic and end-systolic volumes (LVEDV and LVESV): absolute values and indexed to body surface area.
   3. Assessment of regional wall motion abnormalities: wall motion scores for the seventeen myocardial segments and wall motion score index.
   4. Pulsed Doppler mitral inflow: E and A wave velocities, and E/A ratio.
   5. Lateral and medial mitral annular tissue Doppler E', A', and S' wave velocities, lateral and medial E/E' ratios.
   6. Left atrial volume: absolute and indexed to body surface area.
2. 2D Speckle tracking echocardiography (STE) of the left ventricle:

   1. Image acquisition:

      Images will be acquired using the same probe for conventional echocardiography of the Philips machine. Digital loops will be acquired from basal, mid, and apical parasternal short axis views, and apical long-axis, two-chamber and four-chamber views. Frame rates have to be higher than fifty frames per second.
   2. Strain analysis:

   The digitally stored clips will be analyzed offline using TomTec software. For each of the three apical views, the operator manually identifies three points: two on each side of the mitral valve, and a third at the apex of the left ventricle (LV). The software automatically detects the endocardium at end-systole and tracks myocardial motion during the entire cardiac cycle. The software automatically calculates the peak longitudinal and circumferential strain for each individual segment in a seventeen-segment left ventricle model, expressed as bull's eye, and calculates global longitudinal / circumferential strain by averaging local strains along the entire left ventricle. The software provides the strain curves for the 16 myocardial segments (excluding the apical cap). Using a similar process for the short axis views, the software automatically detects the endocardium and generates peak radial strain for each myocardial segment.
3. 3D Speckle tracking echocardiography (STE) of the left ventricle:

   1. Image acquisition:

      • Three-dimensional echocardiography Images will be acquired using the same probe of the Philips machine for conventional echocardiography. Images will be acquired from the apical window, taking care to include the entire LV cavity within the pyramidal scan volume. The dataset will be acquired over 4 consecutive cardiac cycles during a short breath-hold to avoid stitching artifacts.
   2. Strain analysis:

      * Offline analysis of global and regional longitudinal, circumferential, and radial strain will be performed using TomTec software.

Cardiac Magnetic Resonance protocol:

Studies will be performed on a 1.5 T unit (AERA [Siemens Medical System, Erlangen, Germany]) using electrocardiographic triggering and a cardiac-dedicated phase-array coil. For the assessment of LV volumes and function, steady-state free precession breath-held cine images (bSSFP) will be acquired in the following orientations: vertical long axis, horizontal long axis and short axis. Standard parameters are: repetition time/echo time 3.6/1.8 ms; flip angle 50-70°; slice thickness 6 mm; matrix 160 × 256; field of view 350-400 mm; and temporal resolution 25 msec. The set of short axis images will encompass the left ventricle entirely, with a between slices gap of 2 mm. For delayed enhancement imaging, a dose of 0.15 mL of gadolinium per kilogram of body weight will be administered and images will be acquired 10 minutes after contrast injection. The sequence used will be a segmented inversion recovery gradient-echo pulse sequence using the same image orientations as the cine images. Scan parameters are: TR/TE 4.01/1.25 ms, flip angle 15°, matrix 208 x256, and voxel size 1.6 x 1.3x5 mm3. T1 is adjusted to achieve optimal nulling of myocardial signal.

All images will be analyzed offline using Philips IntelliSpace Portal V8.0 workstation (Philips Healthcare, Best, The Netherlands) for analysis of LV volumes, function, and infarct size.

Feature tracking strain analysis:

This will be performed offline using Segment Medviso software that estimates myocardial strain curves by computing inter-frame deformation fields using a tracking strategy based on non-rigid image registration. Instead of myocardial boundaries tracking only, the method uses the entire image content (i.e. blood pool and entire myocardium) during the optimization process. Circumferential and radial LV myocardial Lagrangian strain are evaluated on short-axis cine SSFP images; longitudinal Lagrangian strain is derived from vertical long-axis ones. First, both endo- and epicardial contours are manually drawn at end diastole in the long and short-axis. Contours are propagated automatically by the software throughout the cardiac cycle generating myocardial strain and strain rate curves, with both global and regional values.28

Infarct size:

This will be determined using the full width at half maximum (FWHM) technique, which uses half the maximal signal within the scar as the threshold. The total final infarct area is expressed as percentage of the LV volume, given by the sum of the volume of hyperenhancement on delayed contrast enhanced images (necrosis/scar) for all slices divided by the sum of the LV myocardial cross-sectional volumes (%LV).

LV volumes, function, and strain analysis will be performed in both the baseline and follow-up CMR study; the final infarct size will be calculated from the follow-up study.

A second follow-up visit will be scheduled at 6 months of the index event to collect the following data on clinical outcome:

1. Mortality (all-cause and cardiac)
2. Recurrent angina assessed by Canadian Cardiovascular Society (CCS) grading.
3. Re-infarction.
4. Target lesion revascularization (TLR): either repeat percutaneous or surgical revascularization for a lesion anywhere within the stent or the 5-mm borders proximal or distal to the stent.
5. Target vessel revascularization (TVR): Revascularization of the same vessel of the primary event either surgical or percutaneous other than TLR definition.
6. Re-hospitalization for heart failure. Data on compliance to medications will be reported as well. A written informed consent will be obtained from all patient

ELIGIBILITY:
Inclusion Criteria:

* STEMI with time from symptom onset of <48 hours duration.

Exclusion Criteria:

I. Clinical exclusion criteria:

1. STEMI patients receiving fibrinolytic therapy.
2. Cardiogenic shock, clinical, hemodynamic, or electrical instability persisting after primary PCI.
3. History of prior ST elevation myocardial infarction.
4. Unsuccessful angiographic reperfusion (Thrombolysis In Myocardial Infarction [TIMI] flow grade <2).

II. Contraindications to CMR:

1. Cerebral aneurysm clips
2. Cardiovascular implanted electronic devices
3. Electronic implant or device, eg, insulin pump or other infusion pump
4. Cochlear or otologic implant
5. Shunt (spinal or intraventricular)
6. Tissue expander (eg, breast)
7. Metallic foreign body, especially ocular
8. Penile prosthesis.
9. Patients with stage 4 or 5 chronic kidney disease (estimated glomerular filtration rate <30 mL/min/1.73 m2)
10. Known claustrophobia
11. Known/possible pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will enroll 100 consecutive patients with acute STEMI presenting to Aswan Heart Centre catheterization-lab for primary PCI matching the selection criteria. Diagnosis of STEMI will be based upon:
  Sustained ST-segment elevation of at least 1 mm in at least 2 contiguous leads or new/presumably new left bundle branch block, plus
  * Typical anginal pain
  * or diagnostic levels of serum cardiac biomarkers
  * or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Comparing the predictive ability of 2D, 3D speckle tracking echo and feature tracking CMR for adverse remodeling and final infarct size after STEMI | six months
  Determine the predictors of adverse LV remodeling and final infarct size as assessed by strain analysis using 2D and 3D STE and FT-CMR in STEMI patients treated with primary PCI

SECONDARY OUTCOMES:
Determine the additive value of strain analysis over LV ejection fraction and final infarct size in prediction of clinical outcomes | six months
  Determine the additive value of strain analysis to the well-established prognostic value of LV ejection fraction and final infarct size in prediction of clinical outcomes, including major adverse cardiac events within 6 months follow up of the index event.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan Heart Centre, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided